CLINICAL TRIAL: NCT03475446
Title: Modulating the Effect of a Computerized Cognitive Training With Transcranial Electrical Stimulation in Individuals With and Without Memory Impairment
Brief Title: The Effect of tES on a Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-02056
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Memory Impairment
Keywords: Cognitive Training; Memory Impairment; Mild Cognitive Impairment; Alzheimer's Disease; tES; tACS; tDCS
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants are allocated to one of 3 groups: real tACS, real tDCS or sham. Each participant belongs also to a subpopulation with or without memory impairment (Healthy elderly, MCI, AD)
Who Masked: Participant, Investigator
Masking Description: Double blind design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- sham tES healthy elderly (Placebo Comparator): 30 s of sham transcranial electric current stimulation applied via 5x7 cm and 10x10 cm rubber electrodes over the left DLPFC and supraorbital region. Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for 20 minutes.
  Interventions: Device: sham tES healthy elderly
- sham tES MCI (Placebo Comparator): 30 s of sham transcranial electric current stimulation applied via 5x7 cm and 10x10 cm rubber electrodes over the left DLPFC and supraorbital region. Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for 20 minutes.
  Interventions: Device: sham tES MCI
- sham tES AD (Placebo Comparator): 30 s of sham transcranial electric current stimulation applied via 5x7 cm and 10x10 cm rubber electrodes over the left DLPFC and supraorbital region. Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for 20 minutes.
  Interventions: Device: sham tES AD
- real anodal tDCS healthy elderly (Experimental): 20 min of 2 mA real anodal transcranial direct current stimulation applied via 5x7 cm rubber electrode over the left DLPFC and cathodal 10x10 rubber electrode over supraorbital region. Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real anodal tDCS healthy elderly
- real anodal tDCS MCI (Experimental): 20 min of 2 mA real anodal transcranial direct current stimulation applied via 5x7 cm rubber electrode over the left DLPFC and cathodal 10x10 rubber electrode over supraorbital region. Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real anodal tDCS MCI
- real anodal tDCS AD (Experimental): 20 min of 2 mA real anodal transcranial direct current stimulation applied via 5x7 cm rubber electrode over the left DLPFC and cathodal 10x10 rubber electrode over supraorbital region. Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real anodal tDCS AD
- real tACS healthy elderly (Experimental): 20 min of 1 mA real transcranial alternating current stimulation in theta frequency applied via 5x7 cm rubber electrode over the left DLPFC and cathodal 10x10 rubber electrode over supraorbital region. Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real tACS healthy elderly
- real tACS MCI (Experimental): 20 min of 1 mA real transcranial alternating current stimulation in theta frequency applied via 5x7 cm rubber electrode over the left DLPFC and cathodal 10x10 rubber electrode over supraorbital region. Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real tACS MCI
- real tACS AD (Experimental): 20 min of 1 mA real transcranial alternating current stimulation in theta frequency applied via 5x7 cm rubber electrode over the left DLPFC and cathodal 10x10 rubber electrode over supraorbital region. Additional ramp-up and ramp-down phase of 15 s at the beginning and the end of stimulation.
  Interventions: Device: real tACS AD

INTERVENTIONS:
Device: real anodal tDCS healthy elderly — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the real anodal tDCS in the group of healthy elderly.
  Arms: real anodal tDCS healthy elderly
Device: real tACS healthy elderly — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the real tACS in the group of healthy elderly.
  Arms: real tACS healthy elderly
Device: sham tES healthy elderly — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the sham tES in the group of healthy elderly.
  Arms: sham tES healthy elderly
Device: real anodal tDCS MCI — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the real anodal tDCS in the MCI group.
  Arms: real anodal tDCS MCI
Device: real tACS MCI — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the real tACS in the MCI group.
  Arms: real tACS MCI
Device: sham tES MCI — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the sham tES in the MCI group.
  Arms: sham tES MCI
Device: real anodal tDCS AD — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the real anodal tDCS in the AD group.
  Arms: real anodal tDCS AD
Device: real tACS AD — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the real tACS in the AD group.
  Arms: real tACS AD
Device: sham tES AD — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used for the sham tES in the AD group.
  Arms: sham tES AD

SUMMARY:
The aim of this study is to investigate the effect of a transcranial electrical stimulation (tES) on a cognitive training in healthy elderly and memory impaired participants. In order to assess these effects different memory and attention tasks will be performed before and after the training as well as after 6 and 12 months.

DETAILED DESCRIPTION:
As other studies have shown, transcranial direct current stimulation (tDCS) can improve the outcome of memory tasks in Alzheimer's disease (AD), mild cognitive impairment (MCI) and healthy older adults. Only few studies have investigated the effect of the combination of tDCS and a simultaneous cognitive training and to the investigators' knowledge there is no comparison of tDCS and transcranial alternating current (tACS) effects during a cognitive training or for different populations. With results from this study existing trainings can be optimised. In total 180 participants are planned to be included in this study. This number is based on a g*Power estimation. According to this estimation the study has to include 153 participants. Regarding similar studies the investigators assume a dropout rate of 15% resulting in a total of 180 participants (60 AD patients, 60 MCI patients and 60 healthy older adults) This number should make it possible to find the expected mild effects reported in literature.

A mixed-effects ANOVA model with the between-subjects factor stimulation (tDCS, tACS, sham) and the within-subjects factor time will be computed.

ELIGIBILITY:
Inclusion Criteria:

* Able to give their consent to participate in the study
* Native or fluent German speaker
* Normal or corrected to normal vision and hearing
* Ability to visit the study location for 14 appointments

Exclusion Criteria:

* Acute neurological (other than memory impairment) or psychiatric disorders
* Seizures
* Magnetisable implants
* High dose of psychotropic drugs
* Drug or alcohol abuse
* Participation in another study with investigational drug
* tES in the 2 months preceding or during the present study
* Severe head injuries
* Skin disease
* Caffeine 3 hours prior to training

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Memory | Pre-training (40-0 days before start of training)
  The primary outcome is the change in memory performance.Therefore, changes in the MMS/MoCA score (scores: 0-30, higher scores indicate better functioning of global memory and cognition) and a composite memory score will be assessed. The composite memory score is calculated with the scores of the episodic, prospective and working memory tests.
Memory | Post-training (0-40 days after end of training)
  The primary outcome is the change in memory performance.Therefore, changes in the MMS/MoCA score (scores: 0-30, higher scores indicate better functioning of global memory and cognition) and a composite memory score will be assessed. The composite memory score is calculated with the scores of the episodic, prospective and working memory tests.
Memory | Follow-up 1 (6 months after end of training)
  The primary outcome is the change in memory performance.Therefore, changes in the MMS/MoCA score (scores: 0-30, higher scores indicate better functioning of global memory and cognition) and a composite memory score will be assessed. The composite memory score is calculated with the scores of the episodic, prospective and working memory tests.
Memory | Follow-up 2 (12 months after end of training)
  The primary outcome is the change in memory performance.Therefore, changes in the MMS/MoCA score (scores: 0-30, higher scores indicate better functioning of global memory and cognition) and a composite memory score will be assessed. The composite memory score is calculated with the scores of the episodic, prospective and working memory tests.

SECONDARY OUTCOMES:
Mood | Pre-training (40-0 days before start of training)
  Changes in the subjective measure mood, assessed with questionnaire.
Mood | Post-training (0-40 days after end of training)
  Changes in the subjective measure mood, assessed with questionnaire.
Mood | Follow-up 1 (6 months after end of training)
  Changes in the subjective measure mood, assessed with questionnaire.
Mood | Follow-up 2 (12 months after end of training)
  Changes in the subjective measure mood, assessed with questionnaire.
QOL | Pre-training (40-0 days before start of training)
  Changes in the subjective measure quality of life, assessed with questionnaire.
QOL | Post-training (0-40 days after end of training)
  Changes in the subjective measure quality of life, assessed with questionnaire.
QOL | Follow-up 1 (6 months after end of training)
  Changes in the subjective measure quality of life, assessed with questionnaire.
QOL | Follow-up 2 (12 months after end of training)
  Changes in the subjective measure quality of life, assessed with questionnaire.
AODL | Pre-training (40-0 days before start of training)
  Changes in the subjective measure activities of daily living, assessed with questionnaire.
AODL | Post-training (0-40 days after end of training)
  Changes in the subjective measure activities of daily living, assessed with questionnaire.
AODL | Follow-up 1 (6 months after end of training)
  Changes in the subjective measure activities of daily living, assessed with questionnaire.
AODL | Follow-up 2 (12 months after end of training)
  Changes in the subjective measure activities of daily living, assessed with questionnaire.

OTHER OUTCOMES:
Years of Education | 40-20 days before the start of the training with a questionnaire sent by mail.
  Years of education is a possible predictor of the success of the training and will be assessed once.
Cognitive Reserve | 40-20 days before the start of the training with a questionnaire sent by mail.
  Cognitive reserve is a possible predictor of the success of the training and will be assessed once.
Personality | 40-20 days before the start of the training with a questionnaire sent by mail.
  Personality is a possible predictor of the success of the training and will be assessed once.
Motivation | 30-3 days before the start of the training with a questionnaire in the pre-assessment.
  Motivation is a possible predictor of the success of the training and will be assessed once.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Klöppel, Prof, Principal Investigator — University of Bern
Locations (1):
- Klinik für Alterspsychiatrie und Psychotherapie UPD Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krebs C, Peter J, Brill E, Kloppel S, Brem AK. The moderating effects of sex, age, and education on the outcome of combined cognitive training and transcranial electrical stimulation in older adults. Front Psychol. 2023 Sep 22;14:1243099. doi: 10.3389/fpsyg.2023.1243099. eCollection 2023. PMID 37809311